CLINICAL TRIAL: NCT06541782
Title: Effectiveness of Dyadic Creative Arts Therapies (CAT)-Based Intervention for Improvement of Mother-Child Relationship in Children With Intellectual and Developmental Disabilities: A Mixed Methods RCT
Brief Title: Dyadic Creative Arts Therapies-based Intervention for Children With Intellectual and Developmental Disabilities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Tal-Chen Rabinowitch, Principal Investigator, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3107
Record Dates: First submitted 2024-07-19; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Intellectual Disabilities Global Developmental Delay
Keywords: Music and Play Intervention; Dyadic Intervention; Children with Intellectual and Developmental Disabilities; Playfulness; Parental Playfulness; Mother-Child Relationship
MeSH Terms: conditions — Learning Disabilities; Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: Each participating dyad will be randomized into one of two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dyadic CAT-based Intervention (Experimental): This arm (n=30) will include dyadic CAT-based intervention only.
  Interventions: Behavioral: Dyadic CAT-based Intervention
- Psycho-Educational Parent Counseling (Active Comparator): This arm (n=30) will include psycho-educational parent counseling only.
  Interventions: Behavioral: Psycho-Educational Parent Counseling

INTERVENTIONS:
Behavioral: Dyadic CAT-based Intervention — The experimental dyadic CAT-based intervention will promote mutual sensorimotor play, pretend play, songs, and games among the mother-child dyads while encouraging flexibility, creativity, and enjoyment. This intervention will involve eight weekly 45-minute sessions in the families' homes and will be conducted by trained creative art therapists. The dyadic CAT-based intervention will follow a manualized protocol presenting the goals, principles, and proposed activities for the intervention sessions. It will provide instructions for maintaining intervention fidelity, while allowing flexibility to tailor the meetings to each dyad's strengths and needs. The dyadic CAT-based intervention meetings will be recorded using video camera.
  Arms: Dyadic CAT-based Intervention
Behavioral: Psycho-Educational Parent Counseling — This intervention will involve only mothers and will be conducted by trained parent counselors with experience in working with IDD. This intervention will involve eight weekly 45-minute sessions performed online via Zoom. The psycho-educational parent counseling will follow a protocol presenting the goals, principles, and central issues in parenting a child with IDD to improve the parent-child relationship and address concerns and difficulties related to the child's diagnosis, development, and behavior. It will provide general instructions for maintaining study validity and replication, while allowing flexibility to tailor the intervention to each family's needs.
  Arms: Psycho-Educational Parent Counseling

SUMMARY:
Background: Interactions between parents and children with intellectual and developmental disabilities (IDD) tend to be directive and didactic lacking in playfulness and enjoyment. Recent research has shown that parents of children with IDD who engage in more playful, creative, and enjoyable interactions tend to foster more positive relationships with their children. Early interventions have been shown to enhance parent-child interactions and promote cognitive and socio-emotional development in children with IDD.

Objectives: This mixed-methods randomized controlled trial (RCT) study aims to develop a manualized dyadic Creative-Art-Therapies (CAT)-based intervention for children with IDD and their mothers and assess and explore its effects on the quality of the mother-child interaction and relationship.

Methods: This mixed-methods RCT will investigate and compare two conditions: experimental dyadic CAT-based intervention for children with IDD and their mothers and control psycho-educational counseling intended for mothers only. The sample will consist of sixty dyads of children with IDD between the ages of 3-7 and their mothers, who will be randomly assigned either to experimental or control condition. The experimental group (n=30) will receive 8 weekly individual dyadic CAT-based intervention meetings at their homes and involve both the child and the mother, and the control group (n=30) will receive 8 weekly individual psycho-educational counseling meetings online via Zoom and involve the mother only.

DETAILED DESCRIPTION:
Background:

Play is crucial to children's development and establishing positive parent-child relationships. Children with IDD face substantial developmental delays that often impact their play behaviors, inclining them toward solitary and repetitive play activities while reducing their social interactions. Interactions between parents and children with IDD tend to be directive and didactic lacking in playfulness and enjoyment. Parents of children with IDD who engage in more playful, creative, and enjoyable interactions tend to foster more positive relationships with their children. Early interventions have been shown to enhance parent-child interactions and promote cognitive and socio-emotional development in children with IDD. Thus, this novel intervention may benefit children with IDD and their mothers' interactions and relationships, as well as the children's socio-emotional development and the mothers' well-being. The investigators will develop the dyadic play intervention as part of the study while examining feasibility and intervention fidelity.

Objectives: The objectives of this mixed-methods RCT study are: 1) To develop a manualized dyadic CAT-based intervention for children with IDD and their mothers. 2) To measure the effectiveness of the dyadic CAT-based intervention in improving the quality of the mother-child interaction and increasing the mother's and child's playfulness. 3) To explore the mothers' experience within the intervention and its effect on their playfulness, interactions with their children, and the quality of their relationships.

Methods: A mixed-methods approach will be applied, where quantitative and qualitative data are collected and analyzed in parallel.

Participants: The sample will be composed of 60 dyads of children between the ages of 3-7 diagnosed with IDD and their mothers.

Study Design and Procedures: This is a two-arm RCT that will allocate the participating dyads to one of two conditions: experimental arm of dyadic CAT-based intervention or control arm of psycho-educational parent counseling. All mother-child dyads will participate in a baseline assessment meeting (one week before the first intervention meeting) and a final assessment meeting (one week after the last intervention meeting), each meeting lasting approximately 45 minutes. The assessment meetings will measure the quality of the interactions between children with IDD and their mothers and will be video-recorded.

The experimental arm of dyadic CAT-based dyadic intervention will include eight individual weekly sessions of a mother and a child with a music or drama therapist in their home environment, each session lasting approximately 45 minutes. The intervention will aim to facilitate mutual free-play interactions, promote enjoyment and fun, and enhance the parents' and children's playfulness. The dyadic play intervention will be based on the Creative Arts Therapies as they offer a unique approach to cultivating playfulness, creativity, and self-expression, while employing non-verbal and multi-sensorial techniques, especially suited to the cognitive and verbal skills of children with IDD. As a part of this study, a novel intervention treatment guide will be developed and specifically tailored for the studied population.

The control arm of psycho-educational parent counseling will include eight individual weekly sessions of a mother and a parent counselor, each session lasting approximately 45 minutes. The psycho-educational parent counseling will be performed online via Zoom.

Behavioral tasks and semi-structured interviews will be conducted. Quantitative data will include observational measures of emotional availability (EA), parent-child interpersonal synchrony (IPS), parent's playfulness (via Parent Playfulness scales), and child's playfulness (via Test of Playfulness). Each measure will be collected for each dyad during the assessment meetings at two points of time: before and after the intervention period.

Qualitative data will include interviews with 35% of the mothers who will participate in the dyadic CAT-based intervention, and will be collected following the final assessment meeting and two months after the intervention ends.

ELIGIBILITY:
Inclusion Criteria:

* Children between the age of 3-7
* Children with a prior diagnosis of IDD, or studying in special education nursery schools for children with developmental delays
* The children's mothers

Exclusion Criteria:

* Children with additional primary diagnosis of autism spectrum disorder or cerebral palsy
* Children with additional diagnosis of severe physical disability or serious movement limitations
* Children with additional diagnosis of sensory disorders such as blindness or deafness

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Children - all genders are eligible. Parents - mothers only are eligible.
Enrollment: 60 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mother-Child Emotional Availability | Baseline, Post-intervention (1week after intervention)
  Change in quality of Mother-Child Emotional Availability from baseline to post-intervention. Emotional availability will be assessed from social play without toys task, using Emotional Availability scales which score six sub-scales concerned with emotional regulation in the parent-child dyad: Parent sensitivity (ranging from 1 to 9), parent structuring (ranging from 1 to 5), parent non-intrusiveness (ranging from 1 to 5), parent non-hostility (ranging from 1 to 5), child responsiveness (ranging from 1 to 7), and child involving of parent (ranging from 1 to 7). All scores are averaged into a single emotional availability score for each parent-child dyad, with a higher score signifying an optimal outcome of higher emotional availability.
Mother-Child Interpersonal Synchrony | Baseline, Post-intervention (1week after intervention)
  Change in Mother-Child Interpersonal Synchrony from baseline to post-intervention. Interpersonal synchrony will be measured during mutual movement task, using OpenPose, a multi-person 2D pose estimator, to extract skeletal information from the videos. The positions of the mother and child during the mutual movement task will be examined for coherence and variance using cross-wavelet analysis method, forming an index between 0 and 1 of the degree of interpersonal synchrony between mother and child, with a higher score signifying an optimal outcome of higher interpersonal synchrony.

SECONDARY OUTCOMES:
Mother's Parental Playfulness | Baseline, Post-intervention (1 week after intervention)
  Change in Mother's Parental Playfulness from baseline to post-intervention. Parental playfulness will be assessed from free play and symbolic play tasks using Parental Playfulness scale which score three sub-scales concerned with parental creativity, imagination, and humor while playing with their children: parent's playful behavior, following the child's lead, and peer-like behavior. Each subscale ranges from 1 to 7 and all scores are averaged into a single parental playfulness score, with a higher score signifying an optimal outcome of higher parental playfulness.
Child Playfulness | Baseline, Post-intervention (1 week after intervention)
  Change in Child Playfulness from baseline to post-intervention. Child playfulness will be assessed from free play and symbolic play tasks using Test of Playfulness which scores 30 items concerned with the extent, intensity, and skill of the child at free play. Each item ranges from 1 to 3 and all scores are computed into a single child playfulness score, with a higher score signifying an optimal outcome of higher child playfulness.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No